CLINICAL TRIAL: NCT06978790
Title: Generative Artificial Intelligence Nurse Staffing (GAINS) Study
Brief Title: Generative Artificial Intelligence Nurse Staffing Study
Acronym: GAINS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Principal Investigator, Katie Azama, Assistant Professor, University of Hawaii
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 41775
Record Dates: First submitted 2025-05-01; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Burnout, Healthcare Workers
MeSH Terms: conditions — Burnout, Psychological | interventions — Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Standard staffing practice for float pool nurse and nursing assistants. (Experimental): This arm represents the control or standard of staffing practice to assign float pool nurse and nursing assistants.
  Interventions: Other: Generative Artificial Intelligence Nurse Staffing (GAINS) Intervention
- Arm 2: GAINS intervention applied to float pool nurses (Experimental): Generative Artificial Intelligence Nurse Staffing (GAINS) intervention applied to float pool nurses.
  Interventions: Other: Generative Artificial Intelligence Nurse Staffing (GAINS) Intervention
- Arm 3: GAINS intervention applied to float pool nurses and nursing assistants (Experimental): Generative Artificial Intelligence Nurse Staffing (GAINS) intervention applied to float pool nurses and nursing assistants.
  Interventions: Other: Generative Artificial Intelligence Nurse Staffing (GAINS) Intervention

INTERVENTIONS:
Other: Generative Artificial Intelligence Nurse Staffing (GAINS) Intervention — The Generative Artificial Intelligence intervention is an industrial engineering and nursing-informed innovation developed to optimize team-based staffing of registered nurses and nursing assistants. We anticipate that the GAINS intervention will enhance staffing efficiency, reduces reliance on travel nurses, minimizes overtime costs, and supports nurse well-being by proactively managing workload distribution and reducing burnout. At the core of GAINS is a generative AI model that predicts future unit-level staffing needs using historical staffing patterns, patient turnover (admissions and discharges), and patient acuity scores (based on ICU versus medical/surgical status, physician orders, charge nurse input, and other clinical factors) reflective of workload. Based on the prediction, the intervention dynamically recommends float pool assignments by evaluating staffing gaps across units and optimally deploying available nurses and nursing assistants to where they are most needed.

SUMMARY:
This study is guided by Maslach's Burnout Theory and with Normalization Process Theory supporting the implementation of the GAINS intervention by facilitating its integration into routine system-level practice. In Year 1, the investigative team will collaborate with hospital-based nursing leadership and key stakeholders to identify staffing-specific factors essential for operationalizing the GAINS AI model/intervention. In Year 1, the investigators will also conduct a survey amongst nursing staff to measure baseline burnout. In Year 2, the AI-staffing intervention will be implemented with the medical-surgical nursing float pool team. In Year 3, the investigators will first repeat the nurse burnout survey and second, expand the intervention to include the nursing assistant float pool team. In Year 4, the investigators will conduct the final burnout survey with nurses, assess feasibility of GAINS (target vs. actual staffing- nurses and nursing assistants), and assess preliminary efficacy of GAINS to reduce costs related to staffing. the investigators will compare outcomes at three time points (pre, mid, and post-intervention). Interviews with nurses, nursing assistants, unit nurse managers, and leadership will further explicate the intervention's acceptability, feasibility, and impact on burnout.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses, nursing assistants, or key stakeholders
* Employed by The Queen's Medical Center
* Working at least 24 hours per week
* Position associated with medical-surgical units where float pool nurses work

Exclusion Criteria:

* Employees working less than 24 hours per week at The Queen's Medical Center
* Employees whose roles are not related to medical-surgical units

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Maslach's Burnout Inventory | Up to 2.5 years
  Using Maslach's Burnout Inventory, burnout is the primary outcome measure and will assess burnout (1) at baseline over a time frame of 2 weeks, (2) 12-months after the GAINS intervention is applied to the float pool nurses over a time frame of 2 weeks, and 12-months after the GAINS intervention is applied to the float pool nurses and nursing assistants over a time frame of 2 weeks.
Qualitative Interviews to Evaluate Feasibility, Normalization, and Acceptability of the GAINS Intervention | Up to 3 years
  We will interview 10-20 key stakeholders to collect and analyze qualitative data to evaluate the feasibility, normalization, and acceptability of the GAINS intervention.
  T3here are two phases of the GAINS intervention.
  1. Phase I: GAINS study applied to nurses in Year 2
  2. Phase 2: GAINS study applied to nurses and nursing assistants in Year
  These qualitative interviews will be held in Year 3 after Phase 1 over a 1-month time frame and Year 4 after Phase 2 completion of the study over a 1-month time frame. Interviews will be conducted to gather in-depth feedback on the intervention's feasibility, acceptability, and normalized into nursing practice.

SECONDARY OUTCOMES:
Optimization Staffing Rates [Target staffing rate - Actual staffing rate] | Up to 2 years
  Optimization staffing rates (target staffing rate - actual staffing rate) will be tracked at baseline over a 2-weeks, after Phase 1 over 2-weeks, and at the end of the study over 2-weeks.
Total Cost: Travel Nurse and Nurse Overtime | Up to 2 years
  There are two phases of the GAINS intervention.
  1. Phase I: GAINS study applied to nurses in Year 2.
  2. Phase 2: GAINS study applied to nurses and nursing assistants in Year 3.
  The total cost of travel nurses and nurse overtime will be tracked at baseline over 2-weeks, after Phase 1 is complete over a 2-week time frame, and at the end of Phase 2 over a time frame of 2-weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Katie A Azama, PhD, Principal Investigator — University of Hawaii at Manoa

IPD SHARING:
Plan to Share IPD: No